CLINICAL TRIAL: NCT00014768
Title: Study of Metabolic Effects of Pregnancy in Women With Cystic Fibrosis
Status: Terminated | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Utah (Other)
Other Study IDs: 199/15797; UUSOM-IRB-7922-00
Record Dates: First submitted 2001-04-10; First posted 2001-04-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-03

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Glucose; Insulin; Leucine

STUDY DESIGN:
Observational Model: Natural History

INTERVENTIONS:
Drug: glucose
Drug: insulin
Drug: leucine

SUMMARY:
OBJECTIVES: I. Compare the clinical status of pregnant vs non-pregnant women with cystic fibrosis.

II. Determine glucose tolerance during each trimester of pregnancy in these women.

III. Evaluate peripheral insulin sensitivity in these women. IV. Evaluate whole body protein turnover and hepatic glucose production in these women.

V. Determine resting energy expenditure in these women.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo a glucose tolerance test over 3 hours and a potassium body scan on day 1. Patients undergo an indirect calorimetry over 20 minutes on day 2. Patients receive stable-labeled leucine and stable-labeled glucose IV over 3 hours followed by insulin and glucose IV over 4-4.5 hours on day 2 using the hyperinsulinemic euglycemic clamp technique.

Blood and breath samples are collected to measure glucose tolerance, peripheral insulin sensitivity, and whole body protein turnover. Hepatic glucose production is measured by mass spectrophotometry.

Patients maintain a 3-day food journal before pregnancy, during each trimester, and after pregnancy.

Patients undergo each study during the final 2 weeks of each trimester of pregnancy and then at 6 months post-partum.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of cystic fibrosis (CF) and pregnant OR Age, weight, and body mass index matched non-pregnant CF woman or pregnant non-CF woman
* No infection with Burkholderia cepacia
* FEV1 at least 60%

--Prior/Concurrent Therapy--

* At least 3 weeks since prior corticosteroids

--Patient Characteristics--

* Hepatic: No more than one transaminase level greater than 10% above normal

Other:

Pregnant non-CF controls:

* No cigarette smokers
* No history of gestational diabetes mellitus
* No type 1 or 2 diabetes
* No other chronic illness

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Dana S. Hardin, Study Chair — University of Utah
Locations (1):
- University of Utah School of Medicine, Salt Lake City, Utah, United States